CLINICAL TRIAL: NCT04781439
Title: The Effect of Early Switching From Intravenous to Oral Antibiotics Therapy: a Randomized Control Trial
Brief Title: The Effect of Early Switching From Intravenous to Oral Antibiotics Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gia Dinh People Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 50/CN-HĐĐĐ
Record Dates: First submitted 2021-03-02; First posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Skin and Subcutaneous Tissue Infection
Keywords: effectiveness; antibiotics
MeSH Terms: conditions — Cellulitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- non-switching (No Intervention): control group
- IV-to-PO conversion within 48-72 hours (Experimental): early switching
  Interventions: Procedure: IV-to-PO conversion of antibiotics
- IV-to-PO conversion after 72 hours (Experimental): late switching
  Interventions: Procedure: IV-to-PO conversion of antibiotics

INTERVENTIONS:
Procedure: IV-to-PO conversion of antibiotics — IV-to-PO switching of antibiotics treatment
  Arms: IV-to-PO conversion after 72 hours; IV-to-PO conversion within 48-72 hours

SUMMARY:
To date, many studies showed the great benefits of switching from IV to PO antibiotics in some infectious diseases, especially skin and soft tissue, urinary tract, respiratory tract, gallbladder, and biliary tract infection. Higher level of evidence is necessary to confirm the benefit of early switching protocol in infectious condition management. Therefore, we conducted a clinical trial to investigate the effectiveness and cost of IV-to-PO antibiotic switch therapy in some surgical infection conditions.

DETAILED DESCRIPTION:
Introduction: The benefit of early switching from intravenous (IV) to oral (PO)was raising from the last decade. This randomized clinical trial was to evaluate the effect of early switching from IV to PO antibiotics on the outcome of surgical patients at a public hospital.

Methods: Patients admitted for a therapeutic antibiotic to orthopedic and general surgery conditions were randomly assigned to three groups: control (non-switching), early switching (within 48-72 hours), and late switching (after 72 hours). The rate of effectiveness of each arm, length of hospital stay, length of IV antibiotics, and cost were recorded prospectively.

ELIGIBILITY:
Inclusion Criteria:

* on the second day of IV antibiotic
* no difficulties on taking oral medication
* clinical improvement

Exclusion Criteria:

* n/a

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-09-29 (Actual)

PRIMARY OUTCOMES:
rate of effectiveness | 3 months
  rate of effectiveness of the infection treatment

SECONDARY OUTCOMES:
length of hospital stay | 3 months
  length of hospital stay after starting the antibiotic treatment
length of IV antibiotics | 3 months
  length of IV antibiotics usage
cost of treatment | 3 months
  cost of antibiotics

CONTACTS AND LOCATIONS:
Overall Officials: Dung Nguyen, PhD, Study Director — Gia Dinh People Hospital
Locations (1):
- Gia Dinh people hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No